CLINICAL TRIAL: NCT06742918
Title: To Evaluate the Effect of Berberis Extract (HBR) for the Management of Urinary Tract Infections in Females Measured the Efficacy of HBR, and SBM and Their Combination on Uropathogens to Resolve the Manifestations of UTI in Females
Brief Title: Efficacy of Unani Formulations (HBR and SBM) for Treating Uncomplicated UTIs
Acronym: HBR-SBM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamdard University (Other)
Responsible Party: Principal Investigator, Tabiba Huma Sayeed, Lecturer, Hamdard University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hamdard University, Pakistan
Record Dates: First submitted 2024-05-14; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Urinary Tract Infections; Alternative Medicine; Women Health
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: Group I was given the Tablet HBR (Aqueous extract Berberis), Group II received Syrup SBM (A Unani Formulation), and Group III was given a combination of both. The groups were divided based on the treatment findings to evaluate the efficacy of the medicines, i.e. whether these medicines are effective individually against Uropathogens of in combination.
Who Masked: Participant, Investigator
Masking Description: It is a randomized clinical trial. Participants are the patients who came randomly into the settings and enrolled based on inclusion and exclusion criteria. They are divided into three groups. Group I received Tablet HBR (Aqueous Extract Berberis), Group II received Syrup SBM (a Unani formulation) and Group III received a combination of both.
  Investigator is the researcher of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Syrup SBM (Active Comparator): A Unani formulation which was used since many year to resolve the urinary symptoms, and is described in Unani and Ayurveda Books. This group was designed to observe its antimicrobial effects on Uropathogens
  Interventions: Other: Placebo
- Tablet HBR is Aqueous extract of Berberis. (Experimental): Group II was given Tablet HBR (Aqueous extract Berberis). In a literature search it was found that Berberis was very effective against Uropathogens, especially E.coli.
  Interventions: Other: Placebo
- Group III was given the combination of Tablet HBR and Syrup SBM. (Experimental): The study was designed to identify the efficacy of the combination of the two medicines i.e. Tablet HBR and Syrup SBM, as HBR is a good antimicrobial aqueous extract and Syrup SBM is a very efficacious diuretic medicine. therefore, the combined effects were observed
  Interventions: Other: Placebo
- Placebo (Placebo Comparator): Group IV received placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Placebo was given to the Group IV which was 2 grams of glucose.

SUMMARY:
Based on a huge literature search a gap is found for a complete cure of Urinary Tract Infection (UTI) through the management of traditional antibiotic medicine. Therefore, there is a need to develop a cost-effective, easily available, and more potent drug for the management of UTI.

The objective of the study is as follows.

1. UTI in women is a neglected area in underdeveloped countries due to behavioral factors and zero death ratio in women therefore conduct a clinical study of the Unani formulation to assess the efficacy of the formulation.
2. The prices of allopathic medicines are increasing day by day so the investigator wants to give a cost-effective alternative solution.
3. To explore alternative treatments for Urinary Tract Infections with no or less antimicrobial resistance.

It is a comparative study comparing two formulations in three groups. Participants of Group-I received tablet HBR (HBR group), group-II was given syrup SBM (SBM group) and group-III was given a combination of tablets and syrup (HBR+SBM group) daily twice on an empty stomach for 14 days.

Participants visited the clinic after taking medicine for one week and then the second week.

On the first visit and day 14, patients had their checkups and tests. Hence, the justification for this study is to identify the antimicrobial activity of locally available plant materials and their formulations i.e. HBR and SBM, which have been used in Unani medicine practice for a long. Moreover, conduct a clinical trial for the determination of efficacy and drug resistance of these formulations.

DETAILED DESCRIPTION:
Urinary Tract Infection is one of the most common infections globally, and worldwide about 81% of women are involved with UTI. This occurs most frequently between the ages of 16 to 35 years. About 27% of women with a first episode of UTI record a recurrent within 6 months and 48% within the first year. In uncomplicated UTI, the microorganisms involved are Uropathogenic E.coli, Klebsiella pneumoniae, Staphylococcus saprophyticus, Group B Streptococcus, Pseudomonas aeruginosa, and Staphylococcus aureus in Urinary culture. UTI needs proper diagnosis and prompt management, as if left untreated it can have serious consequences with a chance of progression to chronic disease. Therefore there is a need for an alternative solution for its management especially in developing areas.

The current study was designed as randomized clinical trials of a minimum of 76 female patients, conducted in multi-centers for 14 days, as the disease manifested in acute conditions. The Human Trials were conducted from March 2021 to December 2021. Unani Formulations HBR and SBM were used to treat Uncomplicated Urinary Tract Infections.

Tablet HBR was made as an Aqueous Extract of Berberis roots. the species used here was Berberis aristata. HBR (Aqueous extract of Berberis) is black, having a bitter taste and a pungent smell. It gives Yellowish black/ golden color when dissolved in water.

The ingredients of SBM are as follows:

Cichorium intybus seeds Cichorium intybus Roots Cucumis sativus L Seed Cucumis melo L. Seed Foeniculum vulgare Mill seeds Foeniculum vulgare Mill roots Tribulus terrestris Linn. fruits The Tablets and syrup were made by standard methods described in the literature.

Every registered patient filled out a Case Report Form (CRF) and Temperamental assessment form, each participant then went through the screening for UTI i.e. taking Vitals, Ultrasound KUB (Kidney, Urinary bladder), Blood tests (CBC, Serum Urea, and Serum Creatinine), Urinary Physical Examination, Urine Detail Report (DR) and Urine Culture as baseline investigations.

Patients were randomized to receive test drugs for one week either HBR 1 tablet BD on an empty stomach or syrup SBM 1 tablespoon twice a day on an empty stomach or a combination of both. All females were advised to follow up after one week. After a verbal assessment of the symptoms, another week of medicines was given to the participants. After two weeks of medicines, each participant was tested again for Urine Detailed Report and Urine Culture.

The data was analyzed and assessed by Statistical Package for Social Sciences (SPSS) version 22. It was expressed as the mean ± Standard Deviation (SD), frequency of age groups, ethnic groups, signs and symptoms, temperament, and micro-organisms before and after treatment was assessed. Cross tabulations, Chi-Square was applied for comparison of the variants. Cross-tabulation Pearson's Chi-Square Test analyzed drug compliance. The side effects were observed. A comparison of the cost of the conventional antibiotics and test drugs was done.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 to 70 years have symptoms of UTI.
* Women living in Karachi and the surrounding goth (villages) of Hamdard University came into the study settings.
* Women with pregnancy, Type II Diabetes mellitus, and recurrent UTI.
* Women with every socioeconomic status.
* Females either married or unmarried.
* Women having menopause

Exclusion Criteria:

* Women having chronic renal and liver disease.
* Women who have recently used antibiotics.
* Women with complicated UTIs.
* Women having a menstrual cycle during the checkup.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females having symptoms with UTI
Enrollment: 76 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-09-11 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
The Unani formulations HBR & SBM show significant antibacterial effects against E.coli in UTIs, offering a promising alternative to antibiotics. | 14-days
  The Unani formulation, comprising Tablet HBR (aqueous extract of Berberis) and Syrup SBM, has demonstrated antimicrobial and diuretic properties, particularly against E. coli, the most prevalent uropathogens.
  Literature suggests that HBR exhibits significant antimicrobial activity, while Syrup SBM possesses diuretic properties. This synergistic effect can potentially eliminate microbes from the urinary tract. In light of the growing concern of antimicrobial resistance (AMR) associated with synthetic Allopathic antibiotics, this study aims to investigate the efficacy of Tablet HBR and Syrup SBM as alternative antimicrobial and diuretic agents for uncomplicated urinary tract infections (UTIs).
In clinical response, the combination of HBR & SBM showed an improvement or resolution of signs and symptoms, e.g. resolution of burning micturition, lower abdominal pain, smell in urine, etc. | 14-days
  In the two follow-ups, only the side effect observations found was excessive urination in some patients, otherwise, there was no side effect observed. there was complete improvement or resolution in signs and symptoms observed during and after 14 days of the trials.
The combination of Unani Formulations was estimated Cost effective for the trial period of 14-days in outpatients. | 14-days
  The current market value in the local market of one course of fourth generation Antibiotic costs is very high. The cost of Tablet HBR for one course is nominal, and the combination of both Unani Formulations for one course of treatment also costs low. The high annual costs of conventional UTI medicines are another indicator of the burden they place on society. It was estimated that the Unani formulations would not burden society.

SECONDARY OUTCOMES:
The combination of HBR & SBM showed no side effects observed in the 14-day trial. | 14-days
  After 14 days of acute trial, it was found that there were no major side effects from either the Unani formulations, Tablet HBR, or Syrup SBM. The only minor side effect showed was excessive diuresis in some patients.
Improvement in Blood pressure measurements in some patients. | 14-days
  The combination of HBR & SBM showed a lowering effect on blood pressure in some patients. SBM is a diuretic medicine and due to this effect, Blood pressure is lowered, especially in the summer season.

CONTACTS AND LOCATIONS:
Overall Officials: Tabiba Huma Sayeed Siddiqui, M.Phil, Principal Investigator — Hamdard University
Locations (1):
- Shifa-ul-Mulk Memorial Hospital, Karachi, Sindh, Pakistan